CLINICAL TRIAL: NCT03503149
Title: Molecular Tumor Board at the Center for Personalized Medicine Tübingen: a Prospective Observational Study
Brief Title: Molecular Tumor Board at the Center for Personalized Medicine Tübingen
Acronym: MTB@ZPM
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: ZPM-001
Record Dates: First submitted 2018-03-23; First posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Tumor tissue, blood tisssue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — observational study

SUMMARY:
Molecular Tumor Board at the Center for Personalized Medicine

DETAILED DESCRIPTION:
Molecular Tumor Board at the Center for Personalized Medicine The study objectives are

* To ensure a prospective documentation of all patients who are referred to the Molecular Tumor Board in routine clinical care
* To prospectively ensure the documentation of MTB patients with an emphasis to clinical outcome parameters progression-free survival (PFS), overall survival (OS) and further response assessments (e.g. peripheral immunmonitoring, imaging parameters)
* To prospectively assess patient-reported outcome of MTB patients
* To evaluate compliance to MTB suggestions in routine clinical care

ELIGIBILITY:
Inclusion Criteria:

* Given informed consent ("broad consent" of the University Hospital Tübingen)
* ≥ 18 years of age
* Clinical indication for a referral to Molecular Tumor Board by the treating physician

Exclusion Criteria:

* The MTB assists the referring physician with the interpretation and the use of tumor molecular profiling data for deciding on a therapeutic strategy. Therefore, this board is confined to cancer patients and cannot provide any service for non-cancer patients

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced stages of cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  Progression-free survival

SECONDARY OUTCOMES:
Overall survival | an average of 1 year
  Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Tabatabai, Prof, Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
only within a publication